CLINICAL TRIAL: NCT02608047
Title: Studies on the Pathogen, Vector Control and Clinical Treatment of Dengue Fever in Guangzhou
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou 8th People's Hospital (Other)
Responsible Party: Principal Investigator, Fuchun Zhang, Vice present of hospital, Guangzhou 8th People's Hospital
Other Study IDs: 201508020263
Record Dates: First submitted 2015-10-11; First posted 2015-11-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- dengue patients: Dengue patients confirmed by Non-structural protein and RNA
- Healthy controls: Healthy population without any diseases

SUMMARY:
The purpose of this study is to elucidate the local epidemic problem and epidemiological characters of dengue fever in Guangzhou, to establish diagnostic and treatment standard and clinical treatment system of severe cases to reduce the morbidity and mortality of dengue fever.

DETAILED DESCRIPTION:
To study the epidemiological and pathogenic of dengue virus in Guangzhou, which help to reveal the regular prevalent pattern and the natural epidemic focus of dengue fever. To establish dengue virus sequence database of Guangzhou region, research the biological characteristics and molecular characteristics of dengue fever epidemic strains especially in 2014 in Guangzhou region, to determine the source and variation of this epidemic strains , which finally help to reveal the cause of the pandemic.

To investigate the serum epidemiology of 7800 large groups of people in 12 county-level cities in Guangzhou by stratified random sampling method. It will enrich the research database of the dengue fever serological antibody level survey of people in Guangzhou. After that the investigators could provide a scientific reference for setting up a risk evaluation and implementation of targeted control measures, and also provide reference for analysis of the epidemic situation in other areas.

To study on molecular markers predictive of severe dengue fever and protective immunity after dengue virus infection. The investigators will obtain both serotype-specific and cross-reactive antibodies, which is highly protective neutralizing antibodies. Then the investigators will explore the potential for clinical application about these neutralizing antibodies. The dengue virus were sequenced which caused dengue fever or severe dengue fever in 2014, and do bioinformatics analysis to find the genetic loci which may be responsible for virulence of dengue virus.

To sum up the clinical and laboratory data of dengue fever in 2014, to carry out the research on the diagnosis and treatment of dengue fever, to explore the effectiveness, safety and mechanism of Integrated Chinese and Western medicine treatment for dengue fever patients，to establish of a more perfect system for the diagnosis and treatment of dengue fever in China.

ELIGIBILITY:
Inclusion Criteria:

* Dengue patients confirmed by dengue virus NS1 or RNA

Exclusion Criteria:

* Pregnant women
* Fever diseases caused by other viruses
* Combined bacterial infection
* Without complications such as diabetes and tumor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dengue patients
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
All cause severe dengue | One year

CONTACTS AND LOCATIONS:
Overall Officials: Fuchun Zhang, Principal Investigator — Guangzhou NO 8. people's hospital
Locations (1):
- Guangzhou NO 8. people's hospital, Guangzhou, Guangdong, China